CLINICAL TRIAL: NCT05919771
Title: Effects of Rock Climbing on Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Marymount University (Other)
Responsible Party: Principal Investigator, Julie Ries, Professor, Marymount University
Other Study IDs: 831
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: rock climbing — Vertical ascent of a surface specifically designed to elicit the skills that might be required to scale a naturally occurring rock formation

SUMMARY:
This research study is being conducted to understand the outcomes of participation in the Up ENDing Parkinson's rock climbing program (24 sessions, or twice per week for about 12 weeks) on walking & mobility, hand strength & dexterity, and psychological well-being in individuals with Parkinson's Disease (PD). The rock climbing sessions are administered and supervised by Up ENDing Parkinson's, and are tailored to the skill level of the participant. Participants will answer questionnaires and complete physical performance tests twice, first prior to beginning the sessions and then again after the 24 sessions have been completed.

DETAILED DESCRIPTION:
Parkinson's disease (PD) compromises multiple systems (neurological, musculoskeletal, cardiopulmonary, cognitive) over time, leading to functional decline. Additionally, individuals with PD may experience stressors commonly associated with chronic illness that can negatively impact psychological well-being. Exercise is commonly prescribed for individuals with PD and recently, interventions that are vigorous in nature and community- and performance-based are gaining traction (e.g., dancing, boxing, rock climbing). Despite increasing popularity, the evidence-base for these programs is still developing and far from conclusive. Recommendations are strong for: Community-based exercise, intensive aerobic and resistance training, and external cueing (Osborne et al., 2022). Rock climbing (RC) contains each of these elements and could potentially be a therapeutic intervention for people with PD. Yet little is known about the outcomes of this particular form of organized physical activity programs for this health condition. One such program is the rock climbing experiences offered by the UpENDing Parkinson's Rock Climbing (UEPRC).

The specific aims of this study are to characterize the effects of UEPRC on: 1) mobility and walking; 2) upper extremity (UE) functioning and 3) psychological and social well-being.

Participants will complete 24 rock climbing sessions tailored to their skill levels supervised by UEPRC over approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* Diagnosis of Parkinson's disease
* Hoehn & Yahr score 1-3
* able to speak and read in English;
* able to ambulate at least 10 meters with no assistive device or human assistance

Exclusion Criteria:

* neurological disease diagnosis other than PD;
* uncontrolled cardiovascular, pulmonary, neurological, or metabolic disease which may impact the ability to exercise or in which exercise is contraindicated;
* cognitive or psychiatric impairment precluding informed consent or ability to following instructions;
* pregnancy;
* inability to ambulate 10 meters without assistive device or human assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over the age of 18 with mild-to moderate idiopathic Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Change in Community Mobility and Ambulation | Baseline and at 12 weeks
  Test of specific tasks to be accomplished to walk forward on a level surface safely and efficiently as evidence by the Community Balance and Mobility Scale (CBMS). CBMS is scored from 0-96 with higher scores denoting better performance.

SECONDARY OUTCOMES:
Change in Agility | Baseline and at 12 weeks
  Test of the ability to move forward, laterally, and backward on a level surface safely and efficiently as evidence by the Agility T-Test.
Change in Dexterity | Baseline and at 12 weeks
  This test assesses upper extremity dexterity by assessing the time it takes to remove 9 pegs from a tray and place in peg holes and then remove pegs and place them back in tray as measured by the 9-Hole Peg Test.
Change in Reaction Time | Baseline and at 12 weeks
  This test assesses combined cognitive and physical reaction time to initiate a movement response utilizing colored light stimuli as evidenced by using Blaze Pods.
Change in Apathy | Baseline and at 12 weeks
  This survey addresses lack of emotion, interest, concern, or recognition of goals by measuring levels of participant's interest, motivation, and engagement as evidenced by the Starkstein Apathy Scale. The Starkstein Apathy Scale scores range from 0-42 with higher scores representing greater levels of apathy.
Change in Resilience | Baseline and at 12 weeks
  This survey measures one's ability to thrive in the face of adversity as evidenced by the Connor-Davidson Resilience Scale 25 (CD-RISC-25). CD-RISC-25 scores range from 0-100 with higher scores indicating greater resilience.
Change in Social Adaptation | Baseline and at 12 weeks
  This survey measures motivation and behavior as related to work and hobbies, family and relationships, and social situations as evidenced by the Social Adaptation Self-Evaluation Scale (SAS). SAS scores range from 0-63 with higher scores representing better social adaptation.

OTHER OUTCOMES:
Change in Grip strength | Baseline and at 12 weeks
  Measure of force production in the dominant hand using a hand-held dynamometer. The score is force output in pounds, with higher force output representing greater strength.
Change in Quality of Life across Multiple Dimensions: Perception of difficulty with daily life across 8 dimensions of daily living | Baseline and at 12 weeks
  This survey is a multidimensional survey covering mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort as evidenced by the Parkinson's Disease Questionnaire-39 (PDQ-39). PDQ-39 provides scores from 0-100 in each of the 8 domains listed and an overall Summary Index score from 0-100. Lower scores reflect better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Julie D Ries, PhD, Principal Investigator — Marymount University
Locations (1):
- Marymount University, Arlington, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Osborne JA, Botkin R, Colon-Semenza C, DeAngelis TR, Gallardo OG, Kosakowski H, Martello J, Pradhan S, Rafferty M, Readinger JL, Whitt AL, Ellis TD. Physical Therapist Management of Parkinson Disease: A Clinical Practice Guideline From the American Physical Therapy Association. Phys Ther. 2022 Apr 1;102(4):pzab302. doi: 10.1093/ptj/pzab302. PMID 34963139